CLINICAL TRIAL: NCT04026724
Title: Retrospective Cohort Study on Adjuvant Treatment of Coronary Heart Disease Angina Pectoris With Chinese Patent Medicine
Brief Title: Retrospective Clinical Study on Adjuvant Treatment of Coronary Heart Disease Angina Pectoris With Chinese Patent Medicine
Acronym: RCSCD-TCM
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tianjin University of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Chunquan Yu, Director, Tianjin University of Traditional Chinese Medicine
Other Study IDs: RCSCD-TCM
Record Dates: First submitted 2019-07-13; First posted 2019-07-19 (Actual); Last update posted 2019-07-22 (Actual); Status verified 2019-07

CONDITIONS: Atherosclerotic Heart Disease With Angina Nos

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Exposed group: Chinese patent medicine combined with western medicine routine treatment
  Interventions: Drug: Chinese patent medicine
- Non-exposed group: Western medicine routine treatment

INTERVENTIONS:
Drug: Chinese patent medicine — Shexiang Baoxin Pill, Tongxinluo Capsule, Tongmai Yangxin Pill, Xuefu Zhuyu Capsule, Qishen Yiqi Dropping Pill.
  Groups: Exposed group

SUMMARY:
A retrospective cohort study was performed in patients with angina pectoris who were treated with oral Chinese patent medicine and Western medicine.The hospital's medical record management system was used to collect symptoms of angina pectoris, dose and frequency of nitroglycerin use, clinical biochemical test and imaging examination.To explore the clinical efficacy of Chinese patent medicine in the treatment of coronary heart disease with angina pectoris, and provide reliable data support for its clinical application.

ELIGIBILITY:
Inclusion Criteria:

1. Age 35-75 years old, gender is not limited;
2. Admission time is September 1, 2014 - September 1, 1919;
3. Patients with coronary heart disease and angina pectoris in the Department of Cardiology or Outpatient Department, the diagnosis of angina pectoris meets the diagnostic criteria of Western medicine and the standard of TCM syndrome differentiation;
4. Patients who met the criteria for drug treatment, the exposed group was treated with traditional Chinese medicine combined with Western medicine, and the non-exposed group was treated with Western medicine alone.

Exclusion Criteria:

1. Combined with other heart diseases, neurosis, menopausal syndrome, hyperthyroidism, cervical or vertebral artery type cervical spondylosis, gastro-oesophageal reflux disease or esophageal hiatus hernia may cause chest pain;
2. patients with acute myocardial infarction, heart failure, myocarditis, cardiomyopathy, severe heart valve disease, liver failure or renal failure, malignant tumors and severe metabolic diseases, as well as patients with severe symptoms and uncontrollable angina;
3. Pregnant women, lactating women or women of childbearing age who have birth requirements;
4. Mental patients, or cognitive dysfunction;
5. The investigator believes that there are other situations that are not suitable for the trial.

Ages: 35 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The collaboration network of coronary heart disease research medical units formed by the research group, including the First Affiliated Hospital of Tianjin University of Traditional Chinese Medicine, the Second Affiliated Hospital of Tianjin University of Traditional Chinese Medicine, Tianjin Nankai Hospital, Tianjin Chest Hospital, Tianjin Medical University General Hospital, a total of 5 hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 12400 (Estimated)
Dates: Start 2019-09-01 (Estimated); Primary Completion 2020-03-01 (Estimated); Study Completion 2020-09-01 (Estimated)

PRIMARY OUTCOMES:
Symptoms of angina | one year
Dosage and frequency of use of nitroglycerin | one year
Clinical biochemical indicators test | one year
Film degree exam | one year

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin University of Traditional Chinese Medicine, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Lai Z, Liu Y, Huang M, Li L, Li Z, Su J, Pan G, Li B, Gao S, Yu C. Associations Between Atherosclerosis and Elevated Serum Alkaline Phosphatase in Patients With Coronary Artery Disease in an Inflammatory State. Heart Lung Circ. 2023 Sep;32(9):1096-1106. doi: 10.1016/j.hlc.2023.05.012. Epub 2023 Aug 5. PMID 37550157
- [Derived] Wang J, Huang X, Fu C, Sheng Q, Liu P. Association between triglyceride glucose index, coronary artery calcification and multivessel coronary disease in Chinese patients with acute coronary syndrome. Cardiovasc Diabetol. 2022 Sep 16;21(1):187. doi: 10.1186/s12933-022-01615-4. PMID 36114495
- [Derived] Yu L, Li Z, Yang R, Pan G, Cheng Q, He Y, Liu Y, Liu F, Ma M, Yang T, Wang Y, Su J, Zheng Y, Gao S, Xu Q, Li L, Yu C. Impaired Sensitivity to Thyroid Hormones Is Associated With Elevated Blood Glucose in Coronary Heart Disease. Front Endocrinol (Lausanne). 2022 Jun 15;13:895843. doi: 10.3389/fendo.2022.895843. eCollection 2022. PMID 35784545
- [Derived] Su J, Li Z, Huang M, Wang Y, Yang T, Ma M, Ni T, Pan G, Lai Z, Li C, Li L, Yu C. Triglyceride glucose index for the detection of the severity of coronary artery disease in different glucose metabolic states in patients with coronary heart disease: a RCSCD-TCM study in China. Cardiovasc Diabetol. 2022 Jun 6;21(1):96. doi: 10.1186/s12933-022-01523-7. PMID 35668496